CLINICAL TRIAL: NCT01147887
Title: An Open-Label Study to Assess the Effect of Multiple-Dose JNJ26489112 on the Cytochrome P450 Enzymes Using a 3-Probe Substrate Drug Combination in Healthy Subjects
Brief Title: A Pharmacokinetic and Drug Interaction Study of JNJ-26489112 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CR017176; 26489112MDD1002 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: 26489112; Omeprazole; Tolbutamide
MeSH Terms: interventions — Drug Combinations

ARMS (1):
- 001 (Experimental): Drug combination/ 26489112 On Day 1 and on Day 19 a single oral dose of a drug combination consisting of midazolam (2 mg/mL liquid) tolbutamide (a 500 mg tablet) and omeprazole (a 20 mg capsule) will be taken and on Day 4 through Day 21 a single oral dose of two 26489112 tablets will be taken.
  Interventions: Drug: Drug combination/ 26489112

INTERVENTIONS:
Drug: Drug combination/ 26489112 — On Day 1 and on Day 19, a single, oral dose of a drug combination consisting of midazolam (2 mg/mL liquid), tolbutamide (a 500 mg tablet), and omeprazole (a 20 mg capsule) will be taken and on Day 4 through Day 21, a single oral dose of two 26489112 tablets will be taken.

SUMMARY:
The purpose of this study is to evaluate the effect of 26489112 on the pharmacokinetics (blood levels) of a combination of 3 drugs administered to healthy volunteers.

DETAILED DESCRIPTION:
26489112 is a drug that is being tested to see if it may be useful for a number of indications including major depression. This study will compare the effects of 26489112 administered to healthy volunteers alone or in combination with a mixture of 3 drugs consisting of midazolam (a drug used for reducing anxiety or producing drowsiness or anesthesia before certain medical procedures or surgery), omeprazole (a drug used to treat symptoms of gastroesophageal reflux disease (GERD) or other conditions caused by excess stomach acid), and tolbutamide (a drug used for treating type 2 diabetes mellitus in patients when blood sugar cannot be controlled by diet and exercise alone). Approximately 20 healthy adult volunteers will be enrolled and will be treated with study drug for 22 days. Volunteers will be required to stay overnight at the study center to receive study treatment for 4 nights at the beginning of the study and for 4 nights towards the end of the study. On all other occasions, volunteers will make daily visits to the study center to receive treatment with study drug. Participants will take a combination of 3 drugs (omeprazole 20 mg capsule, tolbutamide 500 mg tablet, and midazolam 2mg/mL liquid) orally (by mouth) or 2 tablets of study drug (2648911) orally with 1 cup of water. Blood samples will be collected from study participants at protocol-specified times during the study to determine the concentration of each of the 4 drugs (26489112, midazolam, omeprazole, and tolbutamide) present in plasma (the colorless fluid portion of blood). In addition, a blood sample will be obtained from all enrolled patients before study drug administration for pharmacogenomics research (research to help identify genetic markers of response, to explain variability in the data, or to address emerging clinical issues). The primary outcome measure is the concentration of midazolam, omeprazole, tolbutamide, and 26489112 in plasma measured by protocol-specified pharmacokinetic parameters at protocol-specified time points on Days 1-4 and Dasy 19-22. Safety will be monitored during the study. Healthy volunteers will receive study drug (26489112) orally (by mouth) in the morning from Day 4 through Day 21.

ELIGIBILITY:
Inclusion Criteria:

* If a woman, must be postmenopausal (no spontaneous menses for at least 2 years), surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control (e.g., intrauterine device, double-barrier method, male partner sterilization) before entry and throughout the study and must have a negative serum beta-human chorionic gonadotropin (hCG) pregnancy test at screening
* If a man, must agree to use an adequate contraception method as deemed appropriate by the investigator (e.g., vasectomy at least 6 months before study entry, double barrier, partner using effective contraception) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Body mass index (BMI
* weight [kg]/height [m]2) between 18 and 30 kg/m2 (inclusive), and body weight not less than 50 kg
* Blood pressure between 90 and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic and results from a 12-lead electrocardiogram (ECG) that are consistent with normal cardiac conduction and function
* Nonsmoker for at least 6 months

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease including current suicidal ideation or behavior, infection, known history of G6PD deficiency, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Known clinically significant ophthalmologic examination results or known ocular deficits, including retinal disorders
* History of clinically significant allergies, known allergy to the study drug or any of the excipients of the formulation, or known allergy to heparin or history of heparin-induced thrombocytopenia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The concentration of midazolam, omeprazole, tolbutamide, and 26489112 in plasma measured by protocol-specified pharmacokinetic parameters | Days 1-4 and Days 19-22

SECONDARY OUTCOMES:
The number of patients with adverse events as a measure of safety. | From screening to the end of the study (Day 22) or at the time of early withdrawal from the study
Results from clinical laboratory tests including blood glucose levels as a measure of safety. | From screening to the end of the study (Day 22) or at the time of early withdrawal from the study
Findings from ECGs and vital sign measurements as a measure of safety. | From screening to the end of the study (Day 22) or at the time of early withdrawal from the study
Findings from physical and neurologic examinations performed as a measure of safety. | From screening to the end of the study (Day 22) or at the time of early withdrawal from the study

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Merksem, Belgium